CLINICAL TRIAL: NCT04222426
Title: Can 89Zr-atezolizumab PET Scan Identify Patients With Metastatic Invasive Lobular Breast Cancer Who Will Respond to Chemotherapy-immune Checkpoint Inhibition?
Brief Title: 89Zr-atezolizumab PET Scan and Lobular Breast Cancer
Acronym: ImaGelato
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Cessation of main trial of which this study was a biomarker imaging side study.
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, C.P. Schroder, principal investigator, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201900180
Record Dates: First submitted 2019-04-23; First posted 2020-01-10 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Lobular Metastatic Breast Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 89Zr-atezolizumab PET scan (Experimental): All patients will undergo two 89Zr-atezolizumab PET scans, one at baseline and one after two doses carboplatin induction treatment. The 89Zr-atezolizumab PET scan will be performed 4 days after tracer injection. Procedures within the ImaGelato study will be completed after the two 89Zr-atezolizumab PET scans, but patients will continue treatment with carboplatin combined with atezolizumab in the GELATO trial.
  Interventions: Other: 89Zr-atezolizumab PET scans

INTERVENTIONS:
Other: 89Zr-atezolizumab PET scans — Patients receive a total amount of 10 mg unlabeled atezolizumab, this will be added to the tracer to prevent rapid clearance during imaging. A labeled dose of 37 Megabequerell (MBq) 89Zr-atezolizumab (±10%; 1 Millicurie) will then be administered. The tracer will be administered intravenously (i.v.). All patients will undergo two 89Zr-atezolizumab PET scans, one at baseline and one after two doses carboplatin induction treatment. After each tracer injection, 89Zr-atezolizumab PET scans will be performed on day 4 (96 ± 6h after tracer administration).

SUMMARY:
The exploratory single center feasibility ImaGelato study is conducted as an imaging side study to the Dutch GELATO trial (Assessing efficacy of carboplatin and atezolizumab in metastatic lobular breast cancer). Ten patients with lobular metastatic breast cancer, who are included in the GELATO trial at the UMCG, are eligible for the ImaGelato study.

All patients will undergo two Zirconium-89 (89Zr)-atezolizumab positron emission tomography (PET) scans, one at baseline and one after two doses carboplatin induction treatment. The 89Zr-atezolizumab PET scan will be performed 4 days after tracer injection. Procedures within the ImaGelato study will be completed after the two 89Zr-atezolizumab PET scans, but patients will continue treatment with carboplatin combined with atezolizumab in the GELATO trial.

ELIGIBILITY:
Inclusion Criteria:

1. A patient must meet the inclusion criteria of the GELATO trial
2. Able to give written informed consent and to comply with the ImaGelato protocol

Exclusion Criteria:

1. Contra-indication for 89Zr-atezolizumab PET scan
2. Any approved anti-cancer therapy, including chemotherapy or hormonal therapy within ≤14 days prior to the first 89Zr-atezolizumab injection. Treatment with any other investigational agent or participation in another clinical trial with therapeutic intent within 28 days prior to the first 89Zr-atezolizumab injection.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Change in tumor uptake between 89Zr-atezolizumab PET scan at baseline and after two carboplatin induction treatments, defined as decline or increase of standardized uptake value | 2 years
  Change in tumor uptake between 89Zr-atezolizumab PET scan at baseline and after two carboplatin induction treatments, defined as decline or increase of standardized uptake value (SUV) of 30% or more, described as per lesion and per patient. For the two different time points we will calculate the SUV for all lesions and patients. Relative decrease or increase in SUV units between different time points will be calculated for all lesions and patients, and recorded as percentage of SUV decrease or increase.

SECONDARY OUTCOMES:
The relation between standardized uptake value (SUV) on 89Zr-atezolizumab PET scan, to response to carboplatin-atezolizumab | 2 years
  Relation of 89Zr-atezolizumab tumor uptake (at baseline, after carboplatin induction, and change between the two scans) per lesion and per patient with response to carboplatin-atezolizumab per lesion and per patient. For the 89Zr-atezolizumab PET scans, uptake will be quantified with SUV units for both time points.
The relation of 89Zr-atezolizumab tumor uptake at baseline and after two courses of carboplatin, with tumor biopsy assessments | 2 years
  Relation of 89Zr-atezolizumab tumor uptake at baseline and after carboplatin induction, with tumor biopsy assessments (for example PD-L1 immunohistochemistry (IHC)). We will investigate whether PD-L1 expression is associated with 89Zr-atezolizumab uptake. The relationship between tumor PD-L1 expression (measured in pre-treatment biopsy and induction treatment biopsy), and 89Zr-atezolizumab tumor uptake will be described.

CONTACTS AND LOCATIONS:
Overall Officials: C. P. Schröder, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands